CLINICAL TRIAL: NCT02553967
Title: Breast Reconstruction and Body Map : Assessment by Functional MRI (REMASCO)
Acronym: REMASCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REMASCO-1503
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: functional Magnetic Resonance Imaging (fMRI); Breast reconstructive surgery; Breast Q questionnaire
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate breast reconstruction (Experimental): * Total mastectomy + immediate reconstructive surgery
  * 6 months after surgery : Functional MRI and questionnaires
  Interventions: Device: Functional MRI
- Secondary breast reconstruction (Experimental): * Within 2 months before surgery : Functional MRI
  * Reconstructive surgery
  * 6 months after surgery : Functional MRI and questionnaires
  Interventions: Device: Functional MRI

INTERVENTIONS:
Device: Functional MRI — Functional MRI

SUMMARY:
Breast reconstruction is an integral part of the management of patients with breast cancer and treated by total mastectomy. The aim of breast reconstruction is to get a satisfying aesthetic and functional result (sensitivity) and that would enable the patient to appropriate the reconstructed breast. Patient satisfaction assessed subjectively by questionnaires would be better in autologous reconstructions than in reconstructions by prosthesis.

The aim of our trial is to use functional MRI (fMRI) as an objective evaluation tool to describe the brain functional changes of sensory projections after immediate or secondary breast reconstruction.

DETAILED DESCRIPTION:
Patients responding criteria for selection and not objecting to participate in this trial will address a quality of life questionnaire at baseline. Then the study procedures differ depending on which group the patient belongs to.

Immediate breast reconstruction group : Six months after surgery (or six months after the implantation of the definitive prosthesis in case of use of a tissue expander), a postoperative fMRI will be performed and patients will be asked to complete a quality of life form and a satisfaction form.

Secondary breast reconstruction group :

* In the two months preceding the surgery, a preoperative fMRI will be performed.
* Six months after surgery (or six months after the implantation of the definitive prosthesis in case of use of a tissue expander), a postoperative fMRI will be performed and patients will be asked to complete a quality of life form and a satisfaction form.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with an indication of unilateral total mastectomy with immediate breast reconstruction for initial breast cancer or recurrence, Or patient undergoing a unilateral secondary breast reconstruction
2. WHO performance status less than or equal to 2
3. Age ≥ 18 years
4. For patients of childbearing age, use of an effective contraceptive method for the duration of the study
5. Patient having been informed and having signed an informed consent form for the study.

Exclusion Criteria:

1. Patient undergoing a breast reconstruction by exclusive lipomodelling
2. Contraindication to MRI : claustrophobia, intra-orbital metallic fragment, pregnancy, cochlear implants, incompatible metallic foreign body such as certain pacemaker and mechanical valves
3. Patient with an indication of preoperative radiotherapy or adjuvant chemotherapy according to regional and/or national standards
4. History of brain surgery
5. History of contralateral breast surgery
6. History of prophylactic total mastectomy
7. Reconstruction techniques using a mixed procedure (autologous + prosthesis)
8. Patient on medication that may alter the BOLD signal in MRI
9. Pregnant or breastfeeding women
10. Patient under tutorship or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
BOLD signal change (difference in intensity and anatomic location) in the regions activated during breast palpation between the reconstructed breast and the non-operated breast. | 6 months

SECONDARY OUTCOMES:
BOLD signal change (difference in intensity and anatomic location) in the regions activated during breast palpation between the breast reconstructed using an autologous flap and a prosthesis. | 6 months
BOLD signal change (difference in intensity and anatomic location) in the regions activated during breast palpation between the reconstructed breast and the mastectomy scar before reconstruction. | 6 months
Topography variation in brain sensory projection area after total mastectomy and breast reconstruction. | 6 months
Satisfaction score and pre and postoperative quality-of-life score (Breast Q) according to a Likert scale. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia REGIS, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No